CLINICAL TRIAL: NCT03049813
Title: Virtual Reality Job Interview Training: An Enhancement to Supported Employment in Severe Mental Illness
Brief Title: Virtual Reality Job Interview Training in Severe Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Thresholds Inc. (Industry); SIMmersion, LLC (Industry); University of Utah (Other)
Responsible Party: Principal Investigator, Matthew Smith, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: R01MH110524-01 (NIH); R01MH110524-01 (NIH)
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Results first posted 2022-11-21 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Depressive Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Depressive Disorder | interventions — Employment, Supported

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Some, but not all, outcomes require masking for the assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Job Interview Training (Experimental): Virtual Reality Job Interview Training
  Interventions: Behavioral: Virtual Reality Job Interview Training
- Supported Employment (Services as Usual) (Other): Supported Employment (Services as Usual)
  Interventions: Other: Supported Employment (Services as Usual)

INTERVENTIONS:
Behavioral: Virtual Reality Job Interview Training — Job interview training using virtual reality software created by SIMmersion, Inc, in addition to standard supported employment services.
  Arms: Virtual Reality Job Interview Training
Other: Supported Employment (Services as Usual) — Standard supported employment services.
  Arms: Supported Employment (Services as Usual)

SUMMARY:
This is a randomized controlled trial to evaluate the community-based effectiveness of virtual reality job interview training (VR-JIT). Northwestern University is partnering with Thresholds Inc. to evaluate the effectiveness of VR-JIT at improving interviewing skills and access to employment. In addition, we will evaluate the cost effectiveness of VR-JIT and the process for implementing VR-JIT at Thresholds.

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 18
2. Diagnosis of any of the following:

   1. Any chronic schizophrenia spectrum disorder, including schizophrenia, schizoaffective disorder, delusional disorder, brief psychotic disorder, schizophreniform disorder, other specified schizophrenia spectrum and related disorder, and unspecified schizophrenia spectrum and related disorders;
   2. Any bipolar spectrum disorder beyond bipolar type I and II to include cyclothymia, other specified bipolar and related disorder, and unspecified bipolar and related disorders;
   3. Any depressive disorder, including disruptive mood dysregulation disorder, major depressive disorder, persistent depressive disorder, other specified depressive disorder, and unspecified depressive disorder;
   4. Posttraumatic stress disorder
3. fluency in English
4. 6th grade reading level
5. Enrolled in Supported Employment/Individual Placement Support (IPS)
6. Active IPS enrollee as indicated by at least 1 contact with his/her Employment Specialist in the past 30 days.
7. Currently unemployed or underemployed
8. Planning to go on interviews within 4 weeks of registration on study.
9. Willing to be video recorded for certain study elements.
10. Must have given signed, informed consent prior to registration on study.

Exclusion Criteria:

1. Documented developmental or learning disability.
2. Medical condition that may compromise cognition (e.g., Parkinson's Disease, Alzheimer's Disease, Huntington's Chorea, Moderate or Greater TBI).
3. Uncorrected vision or hearing problems
4. Active suicidal ideation within the last 30 days with at least some intent to act, with or without a specific plan; this would be reflected in a score of 4 or 5 on the Suicidal Ideation section of the Columbia Suicide Severity Rating Scale (CSSRS)
5. A past suicide attempt within the past 30 days that did not include preparatory acts or behavior, but was defined by a potentially self-injurious act committed with at least some wish to die as a result of the act.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Smith, PhD, Principal Investigator — Northwestern University
Locations (4):
- United States (4):
  - Thresholds Bridge South, Chicago, Illinois
  - Thresholds Ogden, Chicago, Illinois
  - Thresholds Bridge Southwest, Chicago, Illinois
  - Thresholds Bridge West, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Smith MJ, Burke-Miller JK, Bornheimer LA, Ross B, Bell MD, McGurk SR, Mueser KT, Brown A, Prestipino J, Borghani N, Nelson K, Lieberman T, Pashka NJ, Razzano LA, Kallen MA. Psychometric properties of the mock interview rating scale for schizophrenia and other serious mental illnesses. Front Psychiatry. 2023 Apr 27;14:1150307. doi: 10.3389/fpsyt.2023.1150307. eCollection 2023. PMID 37181877

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomized Control Trial Phase: 105 people were enrolled and signed consent forms, but 6 people dropped out of the study before randomization and were not assigned to a group. Therefore, the Randomized Control Trial Phase includes 99 people who signed consent forms and were actually randomized into the study.
  Focus Group Phase: This includes both Thresholds staff focus groups as well as focus groups completed by those who received the intervention in the Randomized Control Trial Phase.
Groups:
- Thresholds Staff: Thresholds Staff members who consented to provide implementation data.
- Focus Group: Focus groups completed by Thresholds staff members and by members of the intervention group who received Virtual Reality Job Interview Training.
Period: Randomized Control Trial Phase
Arm/Group | Supported Employment (Services as Usual) | Virtual Reality Job Interview Training | Thresholds Staff | Focus Group
Started (Signed a consent form) | 38 | 61 | 44 | 0
Completed (Employment Outcomes Obtained by 9-Month Follow-Up) | 36 | 54 | 41 | 0
Not Completed | 2 | 7 | 3 | 0
Not completed — Participant placed in nursing home | 0 | 1 | 0 | 0
Not completed — COVID Quarantine | 2 | 3 | 0 | 0
Not completed — Participant was in another concurrent study | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 3 | 0
Period: Focus Group Phase
Arm/Group | Supported Employment (Services as Usual) | Virtual Reality Job Interview Training | Thresholds Staff | Focus Group
Started | 0 | 0 | 0 | 25
Completed | 0 | 0 | 0 | 25
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Thresholds Staff: Only sex, ethnicity, and race were collected for the Thresholds Staff group.
  Not other baseline data was collected for Thresholds Staff.
- Focus Groups: Baseline data were not collected for the Focus Groups.
- Total: Total of all reporting groups
Arm/Group | Supported Employment (Services as Usual) | Virtual Reality Job Interview Training | Thresholds Staff | Focus Groups | Total
Number analyzed (Participants) | 38 | 61 | 44 | 25 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data were not collected for the Thresholds Group and Focus Groups.
  years
    number analyzed (Participants) | 38 | 61 | 0 | 0 | 99
    (all) | 44.5 (12.8) | 47.4 (12.7) |  |  | 46.3 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Thresholds Staff: n=2 participants elected not to respond to the sex question.
  Focus Groups: Baseline data not collected for this group.
  Participants
    number analyzed (Participants) | 38 | 61 | 42 | 0 | 141
    Female | 15 | 32 | 26 | 0 | 73
    Male | 23 | 29 | 16 | 0 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data were not collected for the Focus Groups.
  Participants
    number analyzed (Participants) | 38 | 61 | 44 | 0 | 143
    Hispanic or Latino | 2 | 7 | 4 |  | 13
    Not Hispanic or Latino | 36 | 54 | 36 |  | 126
    Unknown or Not Reported | 0 | 0 | 4 |  | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Threshold Staff: n=4 participants elected not to respond to the race question.
  Data were not collected for the Focus Groups.
  Participants
    Black, African American: number analyzed (Participants) | 38 | 61 | 40 | 0 | 139
    Black, African American | 26 | 37 | 19 |  | 82
    White: number analyzed (Participants) | 38 | 61 | 44 | 0 | 143
    White | 12 | 21 | 19 |  | 52
    More than one race: number analyzed (Participants) | 38 | 61 | 44 | 0 | 143
    More than one race | 0 | 2 | 1 |  | 3
    Other: number analyzed (Participants) | 38 | 61 | 44 | 0 | 143
    Other | 0 | 1 | 1 |  | 2
Region of Enrollment [Number; unit: participants] — Region of enrollment for Randomized Control Trial Phase only. Population: Region of enrollment for Randomized Control Trial Phase only.
  participants
    United States: number analyzed (Participants) | 38 | 61 | 44 | 0 | 143
    United States | 38 | 61 | 44 |  | 143
Region of Enrollment [Number; unit: participants] — Region of enrollment for Focus Groups Phase only. Population: Region of Enrollment for Focus Group Phase only.
  participants
    United States: number analyzed (Participants) | 0 | 0 | 0 | 25 | 25
    United States |  |  |  | 25 | 25
Years of Education [Mean (Standard Deviation); unit: years] — Population: The following did not answer the question regarding the years of education completed: n=1 for Virtual Reality Job Interview Training group and n=2 for Supported Employment (Services as Usual).
  Data were not collected for the Thresholds Group and Focus Groups.
  years
    number analyzed (Participants) | 36 | 60 | 0 | 0 | 96
    (all) | 12.7 (1.8) | 12.6 (2.2) |  |  | 12.7 (2.1)
Primary Psychiatric Diagnosis [Count of Participants; unit: Participants] — Population: Data were not collected for the Thresholds Group and Focus Groups.
  Participants
    Schizophrenia: number analyzed (Participants) | 38 | 61 | 0 | 0 | 99
    Schizophrenia | 8 | 14 |  |  | 22
    Bipolar Disorder: number analyzed (Participants) | 38 | 61 | 0 | 0 | 99
    Bipolar Disorder | 12 | 15 |  |  | 27
    Major Depressive Disorder: number analyzed (Participants) | 38 | 61 | 0 | 0 | 99
    Major Depressive Disorder | 8 | 23 |  |  | 31
    Schizoaffective Disorder: number analyzed (Participants) | 38 | 61 | 0 | 0 | 99
    Schizoaffective Disorder | 8 | 9 |  |  | 17
    Other: number analyzed (Participants) | 38 | 61 | 0 | 0 | 99
    Other | 1 | 0 |  |  | 1
    Unknown or Not Reported: number analyzed (Participants) | 38 | 61 | 0 | 0 | 99
    Unknown or Not Reported | 1 | 0 |  |  | 1
Brief Psychiatric Rating Scale [Mean (Standard Deviation); unit: units on a scale] — The Brief Psychiatric Rating Scale (BPRS) consists of 18 items and uses a seven-item Likert scale with 1 = "not present", and 7 = "extremely severe". Sum scores can range from 18 to 126. A higher mean score represents more/severe behavioral health symptoms. Population: Data were not collected for the Thresholds Group and Focus Groups.
  units on a scale
    number analyzed (Participants) | 38 | 61 | 0 | 0 | 99
    (all) | 26.4 (7.2) | 24.0 (5.7) |  |  | 24.9 (6.4)
Community Functioning [Mean (Standard Deviation); unit: units on a scale] — As measured by the Specific Levels of Functioning scale. Possible scores range from 30 to 150, with higher scores indicating better functioning. Population: For the Supported Employment (services as usual) group, n=2 has missing data and did not complete the assessment.
  Data were not collected for the Thresholds Group and Focus Groups.
  units on a scale
    number analyzed (Participants) | 36 | 61 | 0 | 0 | 97
    (all) | 127.3 (14.6) | 130.6 (12.2) |  |  | 129.4 (13.2)
Employment History: Had competitive employment in past 2 years [Count of Participants; unit: Participants] — Population: Data were not collected for the Thresholds Group and Focus Groups.
  Participants
    number analyzed (Participants) | 38 | 61 | 0 | 0 | 99
    (all) | 20 | 24 |  |  | 44
Employment History: Ever employed full-time [Count of Participants; unit: Participants] — Population: Data were not collected for the Thresholds Group and Focus Groups.
  Participants
    number analyzed (Participants) | 38 | 61 | 0 | 0 | 99
    (all) | 25 | 44 | 0 |  | 69
Employment History: Ever employed part-time [Count of Participants; unit: Participants] — Population: Data were not collected for the Thresholds Group and Focus Groups.
  Participants
    number analyzed (Participants) | 38 | 61 | 0 | 0 | 99
    (all) | 30 | 50 |  |  | 80
Days in IPS at Baseline [Mean (Standard Deviation); unit: days] — The number of days a participant has been involved with Supported Employment (IPS) at baseline timepoint. Population: Data were not collected for the Thresholds Group and Focus Groups.
  days
    number analyzed (Participants) | 38 | 61 | 0 | 0 | 99
    (all) | 167.9 (189.4) | 118.2 (132.6) |  |  | 138.1 (158.7)
Substance Use [Mean (Standard Deviation); unit: units on a scale] — Substance Use was measured with the Alcohol Use Disorders Identification Test (AUDIT), the range of possible scores is from 0 to 40, where 0 indicates no problems with alcohol, and higher scores indicate more problems with alcohol. DAST-10 was also used to assess substance use; this is a 10 item scale with yes and no questions. A higher score indicates an increased degree of problems related to drug abuse. Scores can range 0 to 10. Population: Data were not collected for the Thresholds Group and Focus Groups.
  units on a scale
    Drug Abuse Screening Test (DAST): number analyzed (Participants) | 38 | 61 | 0 | 0 | 99
    Drug Abuse Screening Test (DAST) | 1.6 (1.2) | 1.4 (1.0) |  |  | 1.5 (1.1)
    Alcohol Use Disorders Identification Test (AUDIT): number analyzed (Participants) | 38 | 61 | 0 | 0 | 99
    Alcohol Use Disorders Identification Test (AUDIT) | 5.3 (7.3) | 3.1 (4.7) |  |  | 4.0 (5.9)
Cognitive ability [Mean (Standard Deviation); unit: T-score] — Cognitive ability was measured with the MATRICS Consensus Cognitive Battery (MCCB). This battery generates T scores for the following domains: processing speed, attention-vigilance, verbal working memory, verbal learning, visual learning, and reasoning/problem solving. Mean scores were created across these six domains to create a total mean score for overall neurocognition. The MCCB also includes a separate T score for social cognition based on the Mayer-Salovey-Caruso Emotional Intelligence Test. Higher scores represent better cognitive ability. (normative mean = 50; standard deviation = 10) Population: Data were not collected for the Thresholds Group and Focus Groups.
  T-score
    Neurocognition: number analyzed (Participants) | 38 | 61 | 0 | 0 | 99
    Neurocognition | 34.2 (10.0) | 34.6 (8.3) |  |  | 34.4 (8.9)
    Social cognition: number analyzed (Participants) | 38 | 61 | 0 | 0 | 99
    Social cognition | 35.2 (14.0) | 37.4 (16.8) |  |  | 36.5 (15.7)

OUTCOME MEASURES:

1. Primary Outcome: Employment Rates
Description: Employment rates at 9-month follow-up visit measured with questionnaire.
Time Frame: 9 month Follow-Up from Randomization Date
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality Job Interview Training | Supported Employment (Services as Usual)
Number analyzed (Participants) | 54 | 36
Participants | 23 | 10
Statistical Analysis 1: Comparison: Virtual Reality Job Interview Training vs Supported Employment (Services as Usual); Test type: Superiority; p = 0.027, Regression, Logistic — One-sided p value; Adjusted for baseline year of study participation, problematic substance use, social cognition, community functioning, and negative symptoms - anergia
Statistical Analysis 2: Comparison: Virtual Reality Job Interview Training vs Supported Employment (Services as Usual); Test type: Superiority; p = 0.0765, Chi-squared — 1-sided p-value

2. Primary Outcome: Time to Employment
Description: We evaluated the number of days between randomization and obtaining employment using a questionnaire administered over phone interviews with the subject and also verifying with Supported Employment (IPS) tracking system.
Time Frame: 9 month Follow-Up from Randomization Date
Population: Time to employment was only reported for those participants who provided that data and who were employed. Not everyone was employed so they would not have a date or a "time to employment" within the analysis. Therefore, this analysis only reports on the 36 people who did get jobs.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Supported Employment (Services as Usual) | Virtual Reality Job Interview Training
Number analyzed (Participants) | 12 | 24
days | 60.6 (57.1) | 101.3 (76.1)
Statistical Analysis 1: Comparison: Supported Employment (Services as Usual) vs Virtual Reality Job Interview Training; Test type: Superiority; p = 0.062, Regression, Cox — One-sided p value; Adjusting for baseline year of study participation, problematic substance use, social cognition, community functioning, and negative symptoms anergia

3. Secondary Outcome: Job Interview Skills
Description: Interviewing skills will be measured using a role-play measure in which subjects act out two job interview scenarios with trained actors. Interviews will be video recorded and scored. An average of the two scenarios at baseline was used to create a single pretest score and an average of the two scenarios at posttest was used to create a single posttest score. The method of assessment is the job interview skills rating scale as measured by the Mock Interview Rating Scale. Possible scores range from 8 to 40, with higher scores indicating better interview skills.
Time Frame: Pretest (Baseline) and Posttest (approximately 3 months after Baseline)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Virtual Reality Job Interview Training | Supported Employment (Services as Usual)
Number analyzed (Participants) | 54 | 36
score on a scale
  Pretest | 24.6 (0.8) | 25.6 (.6)
  Posttest | 24.8 (0.8) | 27.4 (0.6)
Statistical Analysis 1: Comparison: Virtual Reality Job Interview Training vs Supported Employment (Services as Usual); Test type: Superiority; p = 0.006, Regression, Linear — Adjusting for baseline year of study participation, problematic substance use, social cognition, community functioning, negative symptoms - anergia

4. Secondary Outcome: Interview Self-Confidence
Description: Self-reported interview self-confidence. Participants self-reported their confidence in interview skills at pretest and posttest by using a nine-item survey, with items rated on a 7-point scale (1, extremely unskilled, to 7, extremely skilled); total scores were computed across all items. The minimum score is 9 and the maximum score would be 63. Higher scores indicate higher self-confidence in interview skills.
Time Frame: Pretest (Baseline) and Posttest (approximately 3 months after Baseline)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Virtual Reality Job Interview Training | Supported Employment (Services as Usual)
Number analyzed (Participants) | 54 | 36
score on a scale
  Pretest | 43 (1.5) | 43.7 (1.7)
  Posttest | 47.6 (1.6) | 43.8 (1.8)
Statistical Analysis 1: Comparison: Virtual Reality Job Interview Training vs Supported Employment (Services as Usual); Test type: Superiority; p = 0.013, Regression, Linear — Mixed-effects linear regression models. Covariates include: baseline year, problematic substance use, social cognition, community functioning, and negative symptoms (anergia). One-sided p value

5. Secondary Outcome: Interview Anxiety
Description: Self-reported measure of interviewing anxiety completed at pretest and posttest. Participants rated their interview anxiety with an adapted version of the 34-item Personal Report of Public Speaking Apprehension (PRSPA); the phrase "publics peaking" was replaced with "job interviewing." Items were coded from 1, strongly disagree, to 5, strongly agree. Total scores were computed by using the PRSPA's validated two-step total score procedure with the minimum score being 34 and maximum score being 170. Higher scores indicate higher interview anxiety.
Time Frame: Pretest (Baseline) and Posttest (approximately 3 months after Baseline)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Virtual Reality Job Interview Training | Supported Employment (Services as Usual)
Number analyzed (Participants) | 54 | 36
score on a scale
  Pretest | 100.2 (3.6) | 90.5 (4.5)
  Posttest | 90.4 (3.8) | 88.9 (4.6)
Statistical Analysis 1: Comparison: Virtual Reality Job Interview Training vs Supported Employment (Services as Usual); Test type: Superiority; p = 0.019, Regression, Linear — Mixed-effects linear regression models. Covariates include: baseline year, problematic substance use, social cognition, community functioning, and negative symptoms (anergia). One sided p-value

6. Secondary Outcome: Social Competence
Description: Measured by Social Skills Performance Assessment (SSPA). Roleplay performance: The SSPA includes two brief (3-minute) roleplays in which participants engage in a conversation with an unknown confederate who plays the role of a new neighbor(NN) or a landlord (LL). The NN and LL role plays were video recorded at the pre- and posttest visits and were blindly rated by use of an anchoring system. The NN roleplay was scored on eight items via a 5-point scale (e.g., 5,very interested, to 1, very disinterested), and the LL roleplay was scored on nine items via a 5-point scale (e.g., 5,very focused, to 1, very unfocused). The two role-play scores were combined to create one total pretest score and one total posttest score. Sum scores could have a minimum of 17 and maximum of 85. Higher scores indicated better skills.
Time Frame: Pretest (Baseline) and Posttest (approximately 3 months after Baseline)
Population: 96 participants (37 Supported Employment and 59 Virtual Reality Job Interview Training) completed the pretest Social Skills Performance Assessment (SSPA) at baseline. We are missing data on 3 participants due to technical difficulties (no video recording to score) or participants refusing to complete. The total number dropped to 67 participants (27 Supported Employment and 40 Virtual Reality Job Interview Training) at posttest due to participant drop out or non completion of the posttest visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supported Employment (Services as Usual) | Virtual Reality Job Interview Training
Number analyzed (Participants) | 37 | 59
score on a scale
  Pretest | 3.8 (0.6) | 3.7 (0.7)
  Posttest: number analyzed (Participants) | 27 | 40
  Posttest | 4.0 (0.6) | 3.8 (0.7)
Statistical Analysis 1: Comparison: Supported Employment (Services as Usual) vs Virtual Reality Job Interview Training; For this analysis, only participants who completed both pre-test and posttest were included. If someone completed a pre-test SSPA, but not a posttest SSPA, they were not included in the analysis; Test type: Superiority; p = 0.692, Regression, Linear — Mixed-effects linear regression models. Covariates include: baseline year, problematic substance use, social cognition, community functioning, and negative symptoms (anergia)

7. Secondary Outcome: Psychological Distress - Brief Psychiatric Rating Scale
Description: The Brief Psychiatric Rating Scale (BPRS) consists of 18 items and uses a seven-item Likert scale with 1 = "not present", and 7 = "extremely severe". Sum scores can range from 18 to 126. Higher scores indicate more symptoms.
Time Frame: Pretest (Baseline) and 6 Month Follow Up from Randomization Date
Population: For the outcome measure table, 99 participants (38 Supported Employment and 61 Virtual Reality Job Interview Training) completed the pretest Brief Psychiatric (BPRS) at baseline. The total number dropped to 58 participants (25 Supported Employment and 33 Virtual Reality Job Interview Training) at posttest due to participant drop out or non completion of the 6 Month Follow Up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supported Employment (Services as Usual) | Virtual Reality Job Interview Training
Number analyzed (Participants) | 38 | 61
score on a scale
  Pretest BPRS Total | 26.4 (7.2) | 24.0 (5.7)
  6 Month BPRS Total: number analyzed (Participants) | 25 | 33
  6 Month BPRS Total | 24.6 (9.4) | 23.3 (9.2)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through study completion, an average of 12 months.
Arm/Group | Supported Employment (Services as Usual) | Virtual Reality Job Interview Training
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/59
Other Adverse Events (participants affected / at risk) | 0/38 | 0/59

LIMITATIONS AND CAVEATS:
Employment specialists implemented VR-JIT at a central computer lab, which was changed to research staff at local neighborhood sites. Research staff stepped in to avoid delays. Recruitment challenges necessitated reducing targeted enrollment from 160 to 133 participants and from a 1:1 randomization scheme to 3:2 randomization . We initially planned to include only participants who were within 2 weeks of their enrollment in IPS. However, we expanded to all clients currently receiving IPS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT03049813/Prot_SAP_000.pdf
  • Informed Consent Form: RCT Consent Form (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT03049813/ICF_001.pdf
  • Informed Consent Form: Staff Consent Form (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT03049813/ICF_002.pdf
  • Informed Consent Form: Focus Group Consent Form (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT03049813/ICF_003.pdf